CLINICAL TRIAL: NCT03774342
Title: The Influence of Cognitive Decline on Quality of Life After Coronary Bypass
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, I.C.C. van der Horst, Associate professor, University Medical Center Groningen
Other Study IDs: 2018226; 2018/226 (Other: METc - University Medical Center Groningen)
Record Dates: First submitted 2018-10-28; First posted 2018-12-12 (Actual); Last update posted 2019-01-11 (Actual); Status verified 2018-12

CONDITIONS: Coronary Artery Bypass; Cognitive Dysfunction
Keywords: Coronary artery bypass grafting; Quality of life; Cognitive dysfunction; Sarcopenia
MeSH Terms: conditions — Cognitive Dysfunction; Sarcopenia | interventions — Coronary Artery Bypass

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CABG-patients: We will study one group of patients all scheduled for a Coronary Artery Bypass Grafting-procedure. This observational study consists of one group.
  Interventions: Procedure: Coronary Artery Bypass Grafting

INTERVENTIONS:
Procedure: Coronary Artery Bypass Grafting — Patients undergoing coronary artery bypass grafting

SUMMARY:
During the last decades improvements in operative techniques and perioperative care have led to a steady decline in mortality after cardiac surgery. Good survival rates have been shown repeatedly although elderly patients have an increased risk for prolonged hospital stay and postoperative complications such as neurological and pulmonary problems. Post-operative cognitive decline (POCD) is common after cardiac surgery and although this cognitive decline can be subtle, in elderly vulnerable patients even a small decline can have important consequences such as a decreased quality of life and loss of independence. Recent studies among patients after coronary artery bypass grafting (CABG) found that the incidence of POCD varied between 30-60% depending on cognitive tests, time of assessment and patient populations.

Cognitive and physical impairment frequently co-occur in older people. The association between cognitive impairment and functional disability has been investigated in several studies, which demonstrated that cognitive decline is associated with functional disability, also after cardiac surgery. One method for estimation of patients' physical performance is to evaluate sarcopenia. Sarcopenia is defined as a syndrome characterised by progressive and generalised loss of skeletal muscle mass and strength, leading to an increased risk of adverse outcomes such as physical disability, poor quality of life and death. Data on the prevalence of sarcopenia in community-dwelling residents or nursing-homes are widely available, but little is known on (elderly) hospitalized patients after cardiac surgery. The aim of this study is to evaluate the association between post-operative cognitive decline, quality of life (QoL) and sarcopenia in adult patients after coronary artery bypass grafting. The investigators hypothesize that a decreased postoperative QoL is mainly explained by POCD, therefore the primary research question of this study is: What is the influence of post-operative cognitive decline on QoL after CABG? The secondary research question is: Is there an association between postoperative sarcopenia and a decreased postoperative QoL?

DETAILED DESCRIPTION:
Study design:

The investigators will conduct a prospective observational cohort study to evaluate QoL, cognitive decline and sarcopenia in adult patients after coronary artery bypass grafting. The investigators hypothesize that cognitive decline is more associated with QoL than sarcopenia. QoL will be measured using the RAND-36 questionnaire. Cognitive functioning will be measured using several cognitive tests and sarcopenia will be evaluated by measuring muscle mass and muscle strength. The investigators will explore different subgroups according to age including elderly patients (e.g. patients aged 80 years or older at the time of surgery), according to a prolonged stay at the Intensive Care Unit (>24 hours) and according to comorbidities (i.e. diabetes, pulmonary disease, renal failure).

Data collection method:

Routinely, patients planned for CABG are admitted to the cardiothoracic ward one day before surgery. On the day of admittance (one day before surgery) patients will be asked to perform a simple brief battery of 4 computerized tests of cognitive function. At the same time, muscle mass will be assessed using a bioelectrical impedance instrument (BIA) and muscle strength will be assessed using a handgrip strength device. Patients wil also be asked to fill-in a quality of life questionnaire (RAND-36 health survey). Three days after surgery assessments of cognitive functioning, muscle mass and muscle strength will be repeated. Six months after surgery patients will be visited at home where cognitive functioning, muscle strength, muscle mass and QoL will be reassessed.

Study parameters:

1. The primary outcome will be quality of life assessed using the RAND-36 version 2 questionnaire. The questionnaire is widely validated, has a good reliability and includes eight health domains: physical functioning, social functioning, role limitations due to physical health problems, role limitations due to emotional problems, mental health, vitality, pain and general health perception. Outcomes at each dimension will be defined on a scale between 0 and 100; a higher score is equivalent to better health.
2. Cognitive function will be assessed using the brief computerised cognitive test battery (cogstate Ltd, Melbourne, Vic., Australia). This set of tests consists of the detection task, the identification task, the one card learning task and the one back task assessing psychomotor speed, selective attention, visual learning and working memory, respectively. For each postoperative cognitive test, a standardized change in Z-score will be calculated from the difference between the postoperative and baseline score. Of all individual tests the standardized Z-scores will be summed up to generate a composite Z-score. POCD is defined as a Z-score < -2 in two or more individual tasks or a composite Z-score of < -2.
3. To detect sarcopenia the European Working Group on Sarcopenia in Older People (EWGSOP) recommends measurement of both the presence of low muscle mass and low muscle function. Bioelectrical impedance analysis (BIA) can be used for estimation of muscle mass and assessment of handgrip strength can be used for estimation of muscle function.

   * Bio-impedance analysis: BIA estimates the volume of fat and lean body mass. For the calculation of muscle mass we will use the measurements Resistance (RZ), Reactance (Xc) and Phase Angle (Pa) obtained with BIA. These values will be computed by empirically formulated equations based on healthy people with a hydration of the lean body mass around 73%, leading to values for muscle mass (MM), body cell mass (BCM), fat mass (FM) and fat free mas (FFM). Bioelectrical impedance analysis will be performed using a BIA 101 Anniversary edition (AKERN, Florence, Italy). Cut-off values based on normative populations of men and women ≥ 60 years and recommended by the EWGSOP will be used as reference for our study population.
   * Handgrip strength: Muscle strength of the upper extremities will be tested with a hand dynameter measured using the dominant hand. To become familiar with the test, patients will be allowed to perform one practice-test, and then three consecutive tests will be carried out with one minute rest between tests. Only the highest score of the handgrip test will be used for analysis; results will be compared with the reference values recommended by the EWGSOP guidelines.

Additional data:

Additionally, routinely collected variables such as prognostic factors at baseline, data on the surgical procedure and the occurrence of postoperative complications will be recorded as well. Baseline demographic data will include age, gender, body mass index, education level, log EuroSCORE I and co-morbidity such as diabetes (oral therapy or insulin dependent diabetes), pulmonary disease (prolonged use of steroids or other lung medication), arterial vascular disease (peripheral or abdominal vascular pathology or operation due to arterial vascular disease, renal disease (a reduced renal function prior to surgery with an estimated Glomerular Filtration rate (eGFR) <60 ml/min/1.73 m2) and ventricular function (left ventricular ejection fraction: good >50%, moderate 30-50% or poor <30%). The log EuroSCORE I is a widely used risk stratification system for adult cardiac surgery patients which estimates a mortality risk for each individual patient. Data on surgical procedures will be obtained and include the number of grafts and use of cardiopulmonary bypass.

Postoperative complications include:

* Delirium during hospital admittance defined as:

  1. A delirium observation scale score ≥ 3 at hospital ward and/or
  2. A positive confusion assessment method (CAM)-ICU score at the ICU and/or
  3. Diagnosis confirmed by a psychiatrist or geriatrist according to the Diagnostic and Statistical Manual (DSM)-IV criteria
* Myocardial infarction (MI) in the postoperative period. Myocardial infarction associated with CABG (within 48 hours after CABG) is arbitrarily defined by elevation of cardiac biomarker values >10 x 99th percentile upper reference limit (URL) in patients with normal baseline cardiac troponin values. In addition, either (I) new pathological Q waves or new LBBB, or (II) angiographic documented new graft or new native coronary artery occlusion, or (III) imaging evidence of new loss of viable myocardium or new regional wall motion abnormality. After 48 hours, the standard definition of myocardial infarction is appropriate. The following criteria meets the diagnosis for MI: detection of a rise and/or fall of cardiac biomarker values, preferably cardiac troponin, with at least one value above the 99th percentile URL and in addition, either (I) symptoms of ischaemia, or (II) new or presumed new significant ST-segment-T wave (ST-T) changes or new left bundle branch block (LBBB), or (III) development of pathological Q waves in the ECG, or (IV) imaging evidence of new loss of viable myocardium or new regional wall motion abnormality or identification of an intracoronary thrombus by angiography or autopsy
* Surgical re-exploration within 30 days after surgery: thoracotomy due to bleeding, cardiac tamponade or graft failure
* Deep wound infection within 30 days after surgery: when deeper tissues are affected (muscle, sternum and mediastinum) and one or more of the following three criteria are met:

  1. surgical drainage or refixation
  2. an organism is isolated from culture of mediastina tissue or fluid
  3. antibiotic treatment because of a sternal wound
* Stroke: an acute neurological event within 72 hours after surgery with focal signs and symptoms and without evidence supporting any alternative explanation. Diagnoses of stroke requires confirmation by a neurologist
* Renal failure within 30 days after surgery when one or more of the following criteria are met:

  1. renal replacement therapy (dialysis or CVVH) which was not present preoperatively
  2. highest postoperative creatinine level > 177 μmol/L and a doubling of the preoperative value (the preoperative creatinine value is the value on which the EuroSCORE is calculated)

Additional outcomes will be, stay at the Intensive Care Unit (in hours) and discharge destination (i.e. home, nursing home or other healthcare facility).

Data management:

Data will be recorded using OpenClinica and transferred for analysis using Statistical Package for the Social Sciences (SPSS) version 22 (IBM, Chicago, IL). All study subjects will receive a unique study subject identification (ID). Only a researcher with "study director" account properties in OpenClinica will be able to link study subject ID to patient number.

Sample size assessment:

The sample size calculation is based on the hypothetical association between postoperative cognitive decline and QoL. Cognitive decline is assumed to be the independent variable and quality of life as the dependent variable. Data from a previous study among CABG-patients demonstrated POCD in 26% of the included patients at three months after surgery. POCD was defined as a Z-score < -2 in two or more individual tasks, or a composite Z-score of < -2, and the standard deviation (SD) for POCD in this study was 7.4. Another study on assessment of QoL after cardiac events including 6384 patients reported standard deviations of 10.3 and 11.0. With a minimal clinical important difference set at 5 points for change in QoL (e.g. the difference between the postoperative and baseline score), a sample size of 123 patients wil be required for a two-tailed test at an α of 0.05 and power of 80% to find an association between POCD and QoL. The investigators plan to include 140 patients to account for missing data. The inclusion will start in October 2018 and is expected to be completed by the end of July 2019.

Data analysis:

Characteristics of patients will be presented as proportions (with percentages) for dichotomous variables and as means (with standard deviations) or medians (with interquartile ranges) for continuous variables depending on normality. Differences between baseline and 3 days and 6 months follow-up of QoL, POCD and sarcopenia will be evaluated using paired t-tests or Wilcoxon signed rank test when appropriate.

Linear regression will be used to evaluate the association between POCD and change in QoL. First, unadjusted univariate regression analyses of POCD, sarcopenia and potential confounders will be conducted. The following comorbidities will be considered as potential confounders: arterial vascular disease, BMI, renal disease, ventricular function. Additionally, the following postoperative complications will also be evaluated as potential confounders: delirium, stroke and surgical re-exploration.

Multivariable linear regression analysis will be used to evaluate the association of cognitive decline with sarcopenia as covariate, while adjusting for confounding factors. Age will be forced into the multivariable model as it is considered a covariate based on literature, and sarcopenia measured by muscle strength (handgrip test) and muscle mass (BIA) will also be forced into the model as these will also be considered covariates. We will use a p < 0.25 threshold for inclusion of potential confounding variables in the multivariable model, which will be constructed using forward stepwise regression by adding blocks of variables. The multivariable model with POCD as independent variable and QoL as dependent variable will be adjusted for sarcopenia, as covariates. Assumptions will be checked using the appropriate tests. All tests will be performed two-sided and variables with p-values of less than 0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* adult patients scheduled for elective, isolated on-pump CABG
* able to stand and walk independently
* able to participate in the online screenings module for cognitive function to reduce the amount of missing data for cognitive function

Exclusion Criteria:

* Pre-existing neurological deficits
* Psychiatric illness
* previous cardiac surgery
* pre-existing muscular diseases or missing extremities
* presence of an Internal Cardioverter Defibrillator (ICD), assist device or pacemaker
* large amounts of metal in or around the body
* inability to read or understand Dutch instructions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing elective coronary artery bypass grafting
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2018-10-10 (Actual); Primary Completion 2020-01-31 (Estimated); Study Completion 2020-01-31 (Estimated)

PRIMARY OUTCOMES:
Change in quality of life | at baseline (one day before surgery) and 6 months after surgery
  Quality of life will be assessed using the RAND-36 version 2 questionnaire, a widely validated questionnaire including eight health domains; physical functioning, social functioning, role limitations due to physical health problems, role limitations due to emotional problems, mental health, vitality, pain and general health perception. Outcomes at each domain will be defined on a scale from a minimum score of 0 to a maximum score of 100. A higher score is equivalent to a better health.
Change in cognitive functioning | Two sets of cognitive tests will be performed on the day before surgery; one practice test and a second test that will be used as a baseline test. Follow-up tests will be performed at 3 days and 6 months after surgery.
  Cognitive function will be assessed using a set of computerised cognitive tests.This set of tests consists of the detection task, the identification task, the one card learning task and the one back task assessing psychomotor speed, selective attention, visual learning and working memory, respectively.

SECONDARY OUTCOMES:
Change in muscle strength | All tests will be performed on the day before surgery, three days after surgery and 6 months after surgery.
  Assessment of handgrip strength using the Baseline LiTE Hydraulic Hand Dynamometer will be assessed for estimation of muscle function. To become familiar with the test, patients will be allowed to perform one practice-test, and then three consecutive tests will be carried out with one minute rest between tests. Only the highest score of the handgrip test will be used for analysis; strength is measured in kilograms and the testresults will be compared with the reference values recommended by the EWGSOP guidelines.
Change in muscle mass | All tests will be performed on the day before surgery, three days after surgery and 6 months after surgery.
  Bioelectrical impedance analysis (BIA) will be used for estimation of muscle mass. For the calculation of muscle mass the measurements Resistance, Reactance and Phase Angle will be obtained with BIA. These values will be computed by empirically formulated equations based on healthy people leading to values for muscle mass, body cell mass, fat mass and fat free mass. Cut-off values based on normative populations of men and women and recommended by the sarcopenia work group (EWGSOP) will be used as reference for the study population.

CONTACTS AND LOCATIONS:
Overall Officials: Massimo A Mariani, MD, PhD, Study Chair — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cloin EC, Noyez L. Changing profile of elderly patients undergoing coronary bypass surgery. Neth Heart J. 2005 Apr;13(4):132-138. PMID 25696472
- [Background] Markou AL, van der Windt A, van Swieten HA, Noyez L. Changes in quality of life, physical activity, and symptomatic status one year after myocardial revascularization for stable angina. Eur J Cardiothorac Surg. 2008 Nov;34(5):1009-15. doi: 10.1016/j.ejcts.2008.08.003. Epub 2008 Sep 7. PMID 18778947
- [Background] van Harten AE, Scheeren TW, Absalom AR. A review of postoperative cognitive dysfunction and neuroinflammation associated with cardiac surgery and anaesthesia. Anaesthesia. 2012 Mar;67(3):280-93. doi: 10.1111/j.1365-2044.2011.07008.x. PMID 22321085
- [Background] Selnes OA, Gottesman RF, Grega MA, Baumgartner WA, Zeger SL, McKhann GM. Cognitive and neurologic outcomes after coronary-artery bypass surgery. N Engl J Med. 2012 Jan 19;366(3):250-7. doi: 10.1056/NEJMra1100109. No abstract available. PMID 22256807
- [Background] Kok WF, van Harten AE, Koene BM, Mariani MA, Koerts J, Tucha O, Absalom AR, Scheeren TW. A pilot study of cerebral tissue oxygenation and postoperative cognitive dysfunction among patients undergoing coronary artery bypass grafting randomised to surgery with or without cardiopulmonary bypass*. Anaesthesia. 2014 Jun;69(6):613-22. doi: 10.1111/anae.12634. Epub 2014 Apr 22. PMID 24750013
- [Background] Auyeung TW, Kwok T, Lee J, Leung PC, Leung J, Woo J. Functional decline in cognitive impairment--the relationship between physical and cognitive function. Neuroepidemiology. 2008;31(3):167-73. doi: 10.1159/000154929. Epub 2008 Sep 11. PMID 18784415
- [Background] Bruce-Keller AJ, Brouillette RM, Tudor-Locke C, Foil HC, Gahan WP, Nye DM, Guillory L, Keller JN. Relationship between cognitive domains, physical performance, and gait in elderly and demented subjects. J Alzheimers Dis. 2012;30(4):899-908. doi: 10.3233/JAD-2012-120025. PMID 22466001
- [Background] Newman MF, Kirchner JL, Phillips-Bute B, Gaver V, Grocott H, Jones RH, Mark DB, Reves JG, Blumenthal JA; Neurological Outcome Research Group and the Cardiothoracic Anesthesiology Research Endeavors Investigators. Longitudinal assessment of neurocognitive function after coronary-artery bypass surgery. N Engl J Med. 2001 Feb 8;344(6):395-402. doi: 10.1056/NEJM200102083440601. PMID 11172175
- [Background] Mathew JP, Podgoreanu MV, Grocott HP, White WD, Morris RW, Stafford-Smith M, Mackensen GB, Rinder CS, Blumenthal JA, Schwinn DA, Newman MF; PEGASUS Investigative Team. Genetic variants in P-selectin and C-reactive protein influence susceptibility to cognitive decline after cardiac surgery. J Am Coll Cardiol. 2007 May 15;49(19):1934-42. doi: 10.1016/j.jacc.2007.01.080. Epub 2007 Apr 30. PMID 17498578
- [Background] Kozora E, Kongs S, Collins JF, Hattler B, Baltz J, Hampton M, Grover FL, Novitzky D, Shroyer AL. Cognitive outcomes after on- versus off-pump coronary artery bypass surgery. Ann Thorac Surg. 2010 Oct;90(4):1134-41. doi: 10.1016/j.athoracsur.2010.05.076. PMID 20868803
- [Background] Goodpaster BH, Park SW, Harris TB, Kritchevsky SB, Nevitt M, Schwartz AV, Simonsick EM, Tylavsky FA, Visser M, Newman AB. The loss of skeletal muscle strength, mass, and quality in older adults: the health, aging and body composition study. J Gerontol A Biol Sci Med Sci. 2006 Oct;61(10):1059-64. doi: 10.1093/gerona/61.10.1059. PMID 17077199
- [Background] Delmonico MJ, Harris TB, Lee JS, Visser M, Nevitt M, Kritchevsky SB, Tylavsky FA, Newman AB; Health, Aging and Body Composition Study. Alternative definitions of sarcopenia, lower extremity performance, and functional impairment with aging in older men and women. J Am Geriatr Soc. 2007 May;55(5):769-74. doi: 10.1111/j.1532-5415.2007.01140.x. PMID 17493199
- [Background] Cruz-Jentoft AJ, Landi F, Schneider SM, Zuniga C, Arai H, Boirie Y, Chen LK, Fielding RA, Martin FC, Michel JP, Sieber C, Stout JR, Studenski SA, Vellas B, Woo J, Zamboni M, Cederholm T. Prevalence of and interventions for sarcopenia in ageing adults: a systematic review. Report of the International Sarcopenia Initiative (EWGSOP and IWGS). Age Ageing. 2014 Nov;43(6):748-59. doi: 10.1093/ageing/afu115. Epub 2014 Sep 21. PMID 25241753
- [Background] Fredrickson J, Maruff P, Woodward M, Moore L, Fredrickson A, Sach J, Darby D. Evaluation of the usability of a brief computerized cognitive screening test in older people for epidemiological studies. Neuroepidemiology. 2010;34(2):65-75. doi: 10.1159/000264823. Epub 2009 Dec 11. PMID 20016215
- [Background] Rasmussen LS, Larsen K, Houx P, Skovgaard LT, Hanning CD, Moller JT; ISPOCD group. The International Study of Postoperative Cognitive Dysfunction. The assessment of postoperative cognitive function. Acta Anaesthesiol Scand. 2001 Mar;45(3):275-89. doi: 10.1034/j.1399-6576.2001.045003275.x. PMID 11207462
- [Background] VanderZee KI, Sanderman R, Heyink JW, de Haes H. Psychometric qualities of the RAND 36-Item Health Survey 1.0: a multidimensional measure of general health status. Int J Behav Med. 1996;3(2):104-22. doi: 10.1207/s15327558ijbm0302_2. No abstract available. PMID 16250758
- [Background] Cruz-Jentoft AJ, Baeyens JP, Bauer JM, Boirie Y, Cederholm T, Landi F, Martin FC, Michel JP, Rolland Y, Schneider SM, Topinkova E, Vandewoude M, Zamboni M; European Working Group on Sarcopenia in Older People. Sarcopenia: European consensus on definition and diagnosis: Report of the European Working Group on Sarcopenia in Older People. Age Ageing. 2010 Jul;39(4):412-23. doi: 10.1093/ageing/afq034. Epub 2010 Apr 13. PMID 20392703
- [Background] Janssen I, Baumgartner RN, Ross R, Rosenberg IH, Roubenoff R. Skeletal muscle cutpoints associated with elevated physical disability risk in older men and women. Am J Epidemiol. 2004 Feb 15;159(4):413-21. doi: 10.1093/aje/kwh058. PMID 14769646
- [Background] Lauretani F, Russo CR, Bandinelli S, Bartali B, Cavazzini C, Di Iorio A, Corsi AM, Rantanen T, Guralnik JM, Ferrucci L. Age-associated changes in skeletal muscles and their effect on mobility: an operational diagnosis of sarcopenia. J Appl Physiol (1985). 2003 Nov;95(5):1851-60. doi: 10.1152/japplphysiol.00246.2003. PMID 14555665
- [Background] Roques F, Michel P, Goldstone AR, Nashef SA. The logistic EuroSCORE. Eur Heart J. 2003 May;24(9):881-2. doi: 10.1016/s0195-668x(02)00799-6. No abstract available. PMID 12727160
- [Background] Thygesen K, Alpert JS, Jaffe AS, Simoons ML, Chaitman BR, White HD; Writing Group on the Joint ESC/ACCF/AHA/WHF Task Force for the Universal Definition of Myocardial Infarction; Thygesen K, Alpert JS, White HD, Jaffe AS, Katus HA, Apple FS, Lindahl B, Morrow DA, Chaitman BA, Clemmensen PM, Johanson P, Hod H, Underwood R, Bax JJ, Bonow RO, Pinto F, Gibbons RJ, Fox KA, Atar D, Newby LK, Galvani M, Hamm CW, Uretsky BF, Steg PG, Wijns W, Bassand JP, Menasche P, Ravkilde J, Ohman EM, Antman EM, Wallentin LC, Armstrong PW, Simoons ML, Januzzi JL, Nieminen MS, Gheorghiade M, Filippatos G, Luepker RV, Fortmann SP, Rosamond WD, Levy D, Wood D, Smith SC, Hu D, Lopez-Sendon JL, Robertson RM, Weaver D, Tendera M, Bove AA, Parkhomenko AN, Vasilieva EJ, Mendis S; ESC Committee for Practice Guidelines (CPG). Third universal definition of myocardial infarction. Eur Heart J. 2012 Oct;33(20):2551-67. doi: 10.1093/eurheartj/ehs184. Epub 2012 Aug 24. No abstract available. PMID 22922414
- [Background] Sacco RL, Kasner SE, Broderick JP, Caplan LR, Connors JJ, Culebras A, Elkind MS, George MG, Hamdan AD, Higashida RT, Hoh BL, Janis LS, Kase CS, Kleindorfer DO, Lee JM, Moseley ME, Peterson ED, Turan TN, Valderrama AL, Vinters HV; American Heart Association Stroke Council, Council on Cardiovascular Surgery and Anesthesia; Council on Cardiovascular Radiology and Intervention; Council on Cardiovascular and Stroke Nursing; Council on Epidemiology and Prevention; Council on Peripheral Vascular Disease; Council on Nutrition, Physical Activity and Metabolism. An updated definition of stroke for the 21st century: a statement for healthcare professionals from the American Heart Association/American Stroke Association. Stroke. 2013 Jul;44(7):2064-89. doi: 10.1161/STR.0b013e318296aeca. Epub 2013 May 7. PMID 23652265
- [Background] Oldridge N, Hofer S, McGee H, Conroy R, Doyle F, Saner H; (for the HeartQoL Project Investigators). The HeartQoL: Part I. Development of a new core health-related quality of life questionnaire for patients with ischemic heart disease. Eur J Prev Cardiol. 2014 Jan;21(1):90-7. doi: 10.1177/2047487312450544. Epub 2012 Jul 20. PMID 22822179
- [Background] Fabrication Enterprises. Baseline LiTE Hydraulic Hand Dynamometer User Manual (1993). www.FabricationEnterprises.com
- [Derived] Hartog J, Dijkstra S, Dieperink W, Hoekstra T, Fleer J, van der Woude LHV, van der Harst P, Nijsten M, Mariani MA, Blokzijl F. Muscle strength trajectories and their association with postoperative health-related quality of life in patients undergoing coronary artery bypass grafting surgery: a prospective cohort study. BMC Cardiovasc Disord. 2023 Jan 16;23(1):20. doi: 10.1186/s12872-023-03056-7. PMID 36646994
- [Derived] Blokzijl F, Keus F, Houterman S, Dieperink W, van der Horst ICC, Reneman MF, Absalom AR, Mariani MA. Does postoperative cognitive decline after coronary bypass affect quality of life? Open Heart. 2021 Apr;8(1):e001569. doi: 10.1136/openhrt-2020-001569. PMID 33888591